CLINICAL TRIAL: NCT05236517
Title: The Effect of Oral Semaglutide 50 mg Once-daily on Energy Intake, Gastric Emptying, Appetite, Control of Eating and Pharmacokinetics in Participants With Obesity
Brief Title: A Research Study Looking at How 50 mg Semaglutide Daily Affects Food Intake and Emptying of the Stomach in People With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9932-4873; 2021-003341-38 (EudraCT Number); U1111-1266-4375 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-02-04; First posted 2022-02-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: Semaglutide D Dose 1; Drug: Semaglutide D Dose 2; Drug: Semaglutide D Dose 3; Drug: Semaglutide C Dose 4; Drug: Semaglutide C Dose 5 (50 mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Semaglutide C); Drug: Placebo ( Semaglutide D)

INTERVENTIONS:
Drug: Semaglutide D Dose 1 — Tablet given orally
  Arms: Semaglutide
Drug: Semaglutide D Dose 2 — Tablet given orally
  Arms: Semaglutide
Drug: Semaglutide D Dose 3 — Tablet given orally
  Arms: Semaglutide
Drug: Semaglutide C Dose 4 — Tablet given orally
  Arms: Semaglutide
Drug: Semaglutide C Dose 5 (50 mg) — Tablet given orally
  Arms: Semaglutide
Drug: Placebo (Semaglutide C) — Tablet given orally
  Arms: Placebo
Drug: Placebo ( Semaglutide D) — Tablet given orally
  Arms: Placebo

SUMMARY:
This study tests if semaglutide tablets of 50 mg can help people with obesity to lower their food intake compared to placebo. This study also tests how semaglutide 50 mg works on appetite, control of eating (such as cravings and restraints) and how long time the food stays in the stomach after a meal.

In addition, how much semaglutide is in the blood will also be tested. Participants will either get semaglutide or placebo - which treatment participants will get is decided by chance. Participants will receive one semaglutide (or placebo) tablet per day during the 20-week treatment period. The dose of semaglutide is slowly increased every 4 weeks during the study to reach the treatment dose of 50 mg semaglutide taken for 4 weeks.

The study lasts for up to 29 weeks for each person and includes a screening period (up to 4 weeks), a treatment period (20 weeks) and a follow-up period (total of 5 weeks after the last dosing). Participants will have 12 visits with the study doctors at the institute.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years (both inclusive) at the time of signing informed consent
* Body mass index between 30.0 and 45.0 kilogram per meter square (kg/m^2) (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method
* Any disorder which in the investigator's opinion might jeopardise participant safety or compliance with the protocol
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, or endocrinological conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Relative change in energy intake during ad libitum lunch | Baseline to Day 140
  Measured in Percentage

SECONDARY OUTCOMES:
Change in energy intake during ad libitum lunch | Baseline to Day 140
  Measured in kJ
Change in amount of food consumed during ad libitum lunch | Baseline to Day 140
  Measured in g
Change in body weight | Baseline to Day 141
  Measured in Percentage
AUC0-5h,para | 0-5h after standardised meal, Day 141
  Measured in h*μg/mL
AUC0-1h,para | 0-1h after standardised meal, Day 141
  Measured in h*μg/mL
Cmax,para | 0-5h after standardised meal, Day 141
  Measured in μg/mL
tmax,para | 0-5h after standardised meal, Day 141
  Measured in h
Mean postprandial rating - hunger | Day 140
  Measured in mm
Mean postprandial rating - fullness | Day 140
  Measured in mm
Mean postprandial rating - satiety | Day 140
  Measured in mm
Mean postprandial rating - prospective food consumption | Day 140
  Measured in mm
Mean postprandial rating - overall appetite score (OAS) | Day 140
  Measured in mm
Food cravings assessed by Control of Eating Questionnaire (COEQ) | Day 139
  Measured in mm
AUC0-24h,sema,50mg,ss area under these semaglutide-time curve (0-24h) during a dosing interval at steady state | Day 140 to 141
  Measured in nmol*h/L
Cmax,sema,50mg,ss maximum concentration at steady state of semaglutide 50 mg | Day 140 to 175
  Measured in nmol*h/L
tmax,sema,50mg,ss from last dosing to maximum concentration of semaglutide at steady state for semaglutide 50 mg | Day 140 to 175
  Measured in h
t½,sema,50mg,SS terminal half-life of the log concentration time curve | Day 140 to 175
  Measured in h
CL/Fsema,50mg,ss total apparent clearance for semaglutide 50 mg at steady state | Day 140 to 175
  Measured in L/h
Vz/Fsema,50mg,ss apparent volume of distribution during elimination for semaglutide 50 mg at steady state | Day 140 to 175
  Measured in L
Vss/Fsema,50mg,ss apparent volume of distribution at steady state for semaglutide 50 mg | Day 140 to 175
  Measured in L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Gabe MBN, Breitschaft A, Knop FK, Hansen MR, Kirkeby K, Rathor N, Adrian CL. Effect of oral semaglutide on energy intake, appetite, control of eating and gastric emptying in adults living with obesity: A randomized controlled trial. Diabetes Obes Metab. 2024 Oct;26(10):4480-4489. doi: 10.1111/dom.15802. Epub 2024 Jul 31. PMID 39082206